CLINICAL TRIAL: NCT02720432
Title: Early Intervention in Infants With Perinatal Stroke : CIMT Versus HABIT : a Randomized Clinical Trial
Brief Title: Early Intervention in Infants With Perinatal Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1299
Record Dates: First submitted 2016-03-02; First posted 2016-03-25 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Stroke
Keywords: early intervention, infant
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CIMT (Experimental): A soft splint or restraint will be posed to best functioning hand of the infant only during the therapy session. Parents will be educated to perform the therapy, which consists of stimulation of reaching and grasping with the hemiplegic arm.
  The whole intervention period lasts 18 weeks, separated into 3 blocks of 4 weeks intervention and 2 blocks of 3 weeks of rest. During the intervention weeks parents will perform CIMTfor 30 minutes, 6 days a week.
  Interventions: Other: CIMT
- HABIT (Experimental): No restraint will be implemented and instead of promoting unilateral grasping, bimanual grasping will be stimulated. Toys will be precisely selected to stimulate progressed bimanual grasping. The approach of the therapist and parents remain equal.
  The whole intervention period lasts 18 weeks, separated into 3 blocks of 4 weeks intervention and 2 blocks of 3 weeks of rest. During the intervention weeks parents will perform HABIT for 30 minutes, 6 days a week.
  Interventions: Other: HABIT
- Baby-massage (Sham Comparator): 3 sessions of baby-massage will be given by a qualified instructor
  Interventions: Other: baby-massage

INTERVENTIONS:
Other: CIMT — Constraint-induced movement therapy
  Arms: CIMT
Other: HABIT — hand-arm bimanual intensive training
  Arms: HABIT
Other: baby-massage — instructions for baby-massage
  Arms: Baby-massage

SUMMARY:
This current study proposes to analyze the feasibility and effects of the two most used therapies, constraint-induced movement therapy and hand-arm bimanual intensive training, in very young infants (less than one year) with perinatal stroke and with a high risk to develop hemiplegic CP.

DETAILED DESCRIPTION:
Perinatal stroke constitutes an acute presentation of encephalopathy; manifesting as seizure, altered mental status, and/or neurological deficit; between birth and the twenty-eight postnatal day for which a pattern of ischemic brain injury in an arterial distribution is evident by neuroimaging. Following perinatal stroke, approximately 60% of children develop cerebral palsy (usually presenting as spastic hemiplegia), 30-60% experience epilepsy, 25% show language delay, and up to 22% manifest behavioral problems.

The current most predictive tools for early diagnosis of CP are a combination of brain MRI/cUS and a general movements (GM) assessment in the fidgety period (9). Asymmetry of fidgety GMs around 12 weeks post term can be the first clinical signs of hemiplegia.

There are currently two intensive therapy approaches aiming at improving upper limb performance in adults and children (average age 8 years) with established hemiplegic CP: constraint induced movement therapy (CIMT) and Hand-arm bimanual intensive training (HABIT). Those current therapy approaches fundamentally comprise repeated practice of desired movements based on motor learning principles with the adult/ child as an active participant.

Both therapies, in adults and in children with established hemiplegic CP (average age 8 years) are effective and show similar improvements if the dosage of therapy is similar. In contrast, the feasibility and the effects of both therapy approaches at very young age (under age 1 year) is still unknown (22). Exploring these options to treat even before asymmetric hand use has appeared is interesting and promising enough since recent animal studies have demonstrated that there is a critical period of motor system plasticity, and that activity-dependent reorganization of the motor-projection pattern to the hand occurs before about 1 year of age

ELIGIBILITY:
Inclusion Criteria:

* Infants with a perinatal stroke confirmed on neonatal imaging and from who the parents speaks Dutch and live in Belgium, will be included in the study. Only infants showing abnormal 'general movements' between 10 and 15 weeks will be eligible for the intervention part.

Exclusion Criteria:

* Infants with severe genetic abnormalities or malformations, with severe visual impairments or with uncontrolled seizures will be excluded.

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in the score of the Hand assessment for infants (HAI) | before (around 4 months) and after 18 weeks of intervention (around 9 months)
  The HAI is the very new assessment tool to evaluate the hand function and asymmetry in infants age from 2 till 8 months post term.
Change in the score of the Infant motor profile | before (around 4 months) and after 18 weeks of intervention (around 9 months), at one year follow up
  The IMP is a video-based assessment to evaluate the spontaneous motor behavior of infants from 3 months till independent walking around 18 months of age
Change in the score of the Alberta infant motor scale | before (around 4 months) and after 18 weeks of intervention (around 9 months), at one year follow up
  The AIMS is a standardized observational scale to assess the gross motor development from birth till independent walking around 18 months of age.

SECONDARY OUTCOMES:
Bayley scales for infant development-third edition | between 22 and 24 months (2 years)
  The Bayley Scales of Infant and Toddler Development, Third is a validated and extensively used developmental scale for assessing the cognitive, language and motor development from 1 month till 42 months of age.
Parental sense of competence scale | before intervention (around 4months)
  The parenting Sense of Competence scale is a 16-item Likert-scale questionnaire to measure parent's sense of confidence and satisfaction.
Questionnaire satisfaction and impact | after the intervention (around 9 months)
  A questionnaire will be filled out by the parents at the end of the therapy. They will be asked about the satisfaction of the therapy and therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Govaert, Dr, Principal Investigator — Universiteit Gent, vakgroep REVAKI
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No